CLINICAL TRIAL: NCT01143649
Title: Effects of Transcranial DC Stimulation Coupled With Constraint Induced Movement Therapy on Motor Function in Stroke Patients
Brief Title: Use of Transcranial Direct Current Stimulation (tDCS) Coupled With Constraint Induced Movement Therapy in Stroke Patient
Acronym: tdcs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Felipe Fregni, Principal Investigator, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2009p001808
Record Dates: First submitted 2010-04-20; First posted 2010-06-14 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Stroke; Healthy
Keywords: Stroke; Transcranial direct current stimulation; Motor function
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation; Constraint Induced Movement Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- active tDCS + CIMT - stroke patients (Experimental): Participants will receive 5 sessions of tDCS over the primary motor cortex (M1). We will use the following stimulation parameters: intensity of 1mA and for the first 40 minutes of constraint induced movement therapy (CIMT - 10 consecutive sessions Monday- Friday).
  Interventions: Device: transcranial direct current stimulation (tDCS); Procedure: constraint induced movement therapy (CIMT)
- active tDCS + CIMT - Healthy (Experimental): Participants will receive one session of tDCS over the primary motor cortex (M1). We will use the following stimulation parameters: intensity of 1mA and for the first 40 minutes of constraint induced movement therapy (CIMT)
  Interventions: Device: transcranial direct current stimulation (tDCS); Procedure: constraint induced movement therapy (CIMT)
- tACS - Healthy Subjects (Experimental): The investigators will have 40 healthy subjects who will undergo one session of treatment with active tACS (in which the order in which they receive either sham or active transcranial alternating current stimulation (tACS) stimulation will be randomized).
  Interventions: Device: transcranial alternating current stimulation (tACS)
- sham tDCS + CIMT - stroke patients (Sham Comparator): Participants will receive 5 sessions of tDCS over the primary motor cortex (M1). We will use the following stimulation parameters: intensity of 1mA and for the first 40 minutes of constraint induced movement therapy (CIMT - 10 consecutive sessions Monday- Friday). For the sham session, tDCS is turned off after 30seconds.
  Interventions: Device: transcranial direct current stimulation (tDCS); Procedure: constraint induced movement therapy (CIMT)
- sham tDCS + CIMT - Healthy (Sham Comparator): Participants will receive one session of tDCS over the primary motor cortex (M1). We will use the following stimulation parameters: intensity of 1mA and for the first 40 minutes of constraint induced movement therapy (CIMT). The sham stimulation consists of 30 seconds of stimulation at the beginning of the 40 min of treatment.
  Interventions: Device: transcranial direct current stimulation (tDCS); Procedure: constraint induced movement therapy (CIMT)
- sham tACS - Healthy Subjects (Sham Comparator): The investigators will have 40 healthy subjects who will undergo one day of treatment with sham tACS. All participants received active and sham stimulation in a randomized order.
  Interventions: Device: transcranial alternating current stimulation (tACS)

INTERVENTIONS:
Device: transcranial direct current stimulation (tDCS) — Subjects will be stimulated at 1 mA for 40 minutes.
  Arms: active tDCS + CIMT - Healthy; active tDCS + CIMT - stroke patients; sham tDCS + CIMT - Healthy; sham tDCS + CIMT - stroke patients
Procedure: constraint induced movement therapy (CIMT)
  Arms: active tDCS + CIMT - Healthy; active tDCS + CIMT - stroke patients; sham tDCS + CIMT - Healthy; sham tDCS + CIMT - stroke patients
Device: transcranial alternating current stimulation (tACS) — Subjects will be stimulated at 15Hz for 20 minutes.
  Arms: sham tACS - Healthy Subjects; tACS - Healthy Subjects

SUMMARY:
The purpose of this study is to determine whether noninvasive brain stimulation associated with motor learning offers an additional benefit than motor learning alone in patients with stroke.

The investigators hypothesis is that active transcranial direct current stimulation (tDCS) combined with constraint induced movement therapy (CIMT) will induce a greater motor function improvement as compared with sham tDCS combined with CIMT.

DETAILED DESCRIPTION:
In this 3 experiments study we will evaluate the effect of tDCS and constraint induced movement therapy (CIMT) in stroke patients (exp 1) as well as in healthy subjects (control population - exp 2). Finally we will investigate the effect of tACS - transcranial alternating current stimulation - as an alternative to tDCS, on motor function in healthy subjects (exp 3). The two experiments on tDCS are parallels (exp 1 & 2), while the experiment on tACS uses a crossover design (exp 3).

For stroke patients (Exp1), our primary outcome measure is a clinical scale (Jebsen-Taylor Hand Function Test), while for healthy subjects (Exp 2) we investigate the effect of tDCS and CIMIT on cortico-spinal excitability using TMS - transcranial magnetic stimulation. Finally, for the third experiment using tACS, our primary outcome is cortical oscillation, as measured by EEG - electroencephalogram.

ELIGIBILITY:
Inclusion Criteria:

All subjects must be between the ages of 18-90 and must not be pregnant.

Additional Entry criteria for Stroke subject enrollment:

1. First-time clinical ischemic or hemorrhagic cerebrovascular accident - evidenced by a radiological (or physician's) report;
2. Weakness, defined as score of less than 55 (out of 66) on arm motor Fugl-Meyer (FM) scale
3. Stroke onset >6 months prior to study enrollment.

Exclusion Criteria:

1. Significant pre-stroke disability;
2. Major depression, as defined by Hamilton Depression (HAM-D) scale grater then or equal 17 if needed (history of depression before the stroke);
3. Any substantial decrease in alertness, language reception, or attention that might interfere with understanding instructions for motor testing;
4. Excessive pain in any joint of the paretic extremity (not applicable to severe stroke subjects);
5. Contraindications to single pulse Transcranial Magnetic Stimulation (TMS) (TMS will be used to measure cortical excitability) such as metal head implants

   * history of seizures
   * unexplained loss of consciousness
   * metal in the head
   * frequent or severe headaches or neck pain
   * implanted brain medical devices.
6. Contraindications to tDCS

   * metal in the head
   * implanted brain medical devices
7. Advanced liver, kidney, cardiac, or pulmonary disease;
8. A terminal medical diagnosis consistent with survival < 1 year;
9. Coexistent major neurological or psychiatric disease as to decrease number of confounders;
10. A history of significant alcohol or drug abuse in the prior 6 months;
11. Use of carbamazepine and amitriptyline;
12. Subjects may not be actively enrolled in a separate intervention study targeting stroke recovery and
13. Subjects may not have already received constraint induced motor therapy and/or tDCS treatment for stroke;
14. History of epilepsy before stroke (or episodes of seizures within the last six months).
15. Subjects with global aphasia and deficits of comprehension
16. Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2011-04 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Fregni, PhD, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving activities of daily living, and physical and cognitive functioning, in people after stroke. Cochrane Database Syst Rev. 2020 Nov 11;11(11):CD009645. doi: 10.1002/14651858.CD009645.pub4. PMID 33175411

RESULTS

PARTICIPANT FLOW:
Groups:
- tDCS + CIMT - Stroke: Participants will receive tDCS over the primary motor cortex (M1). We will use the following stimulation parameters: intensity of 1mA and for the first 40 minutes of constraint induced movement therapy (CIMT- 10 consecutive sessions Monday- Friday).
  Transcranial Stimulation: Subjects will be stimulated at 1 mA for 40 minutes.
- Sham tDCS + CIMT - Stroke: Participants will receive tDCS over the primary motor cortex (M1). We will use the following stimulation parameters: intensity of 1mA and for the first 40 minutes of constraint induced movement therapy (CIMT- 10 consecutive sessions Monday- Friday).
  Sham stimulation consists of 30secondes of stimulation at the beginning of the 40minutes treatment.
- Healthy Participants: Active tDCS + Motor Training: Each stimulation day will include up to six hours of training termed "shaping" in the non-dominant hand while the dominant hand is restrained in a resting hand splint and secured in a sling. At the start of this training, subjects will undergo 40 minutes of tDCS at 1mA.
- Healthy Participants: Sham tDCS + Motor Training: Each stimulation day will include up to six hours of training termed "shaping" in the non-dominant hand while the dominant hand is restrained in a resting hand splint and secured in a sling. At the start of this training, subjects will undergo 40 minutes of sham tDCS.
- Healthy Participants - Active tACS, Then Sham: Subjects will receive 20 min of active then sham tACS over the primary motor cortex in a randomized order.
- Healthy Participants - Sham tACS, Then Active: Subjects will receive 20 min of sham and then tACS over the primary motor cortex in a randomized order.
Period: Overall Study
Arm/Group | tDCS + CIMT - Stroke | Sham tDCS + CIMT - Stroke | Healthy Participants: Active tDCS + Motor Training | Healthy Participants: Sham tDCS + Motor Training | Healthy Participants - Active tACS, Then Sham | Healthy Participants - Sham tACS, Then Active
Started | 7 | 7 | 10 | 10 | 5 | 5
Completed | 7 | 7 | 10 | 10 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- tDCS + CIMT - Stroke: Participants received active tDCS over the primary motor cortex (M1). We used the following stimulation parameters: intensity of 1mA and for the first 40 minutes of constraint induced movement therapy (CIMT- 10 consecutive sessions Monday- Friday).
  Transcranial Stimulation: Subjects were stimulated at 1 mA for 40 minutes.
- Sham tDCS + CIMT - Stroke: Participants received sham tDCS over the primary motor cortex plus CIMT. The same site and parameters of stimulation were employed, but the stimulator was turned off after 30 seconds of stimulation. This ensured that patients could feel the initial itching sensation at the beginning of tDCS.
- tDCS Active + CIMT - Healthy: Participants received active (1mA - 40min) of the primary motor cortex (M1) bilaterally combined with unilateral motor training and contralateral hand restraint.
- Sham tDCS + CIMT - Healthy: Participants received sham tDCS (1mA - 40min) of the primary motor cortex (M1) bilaterally combined with unilateral motor training and contralateral hand restraint.
- tACS Active&Sham - Healthy: active or sham 15Hz-tACS over of the primary motor cortex (M1) bilaterally.
- Total: Total of all reporting groups
Arm/Group | tDCS + CIMT - Stroke | Sham tDCS + CIMT - Stroke | tDCS Active + CIMT - Healthy | Sham tDCS + CIMT - Healthy | tACS Active&Sham - Healthy | Total
Number analyzed (Participants) | 7 | 7 | 10 | 10 | 10 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 10 | 10 | 10 | 43
  >=65 years | 0 | 1 | 0 | 0 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (12.8) | 50.8 (14.9) | 20.4 (1.7) | 20.4 (1.7) | 35.83 (18.65) | 35.75 (11.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 7 | 7 | 4 | 27
  Male | 3 | 2 | 3 | 3 | 6 | 17

OUTCOME MEASURES:

1. Primary Outcome: Jebsen Taylor Hand Function Test
Description: Jebsen Taylor Hand Function Test: measures hand function in real-life activities, by evaluating the time required to perform 7 different tasks. We used the non-cronstrained hand for the assessments. The sum of the different tasks was used for the analysis.
Time Frame: 2 weeks
Population: The Jebsen Taylor Hand Function Test was only performed in the stroke study (Experiment 1).
Measure: Mean (Standard Error); unit: seconds
Groups:
- tDCS + CIMT: Participants will receive tDCS over the primary motor cortex (M1). We will use the following stimulation parameters: intensity of 1mA and for the first 40 minutes of constraint induced movement therapy (CIMT- 10 consecutive sessions Monday- Friday).
  Transcranial Stimulation: Subjects will be stimulated at 1 mA for 40 minutes.
- Sham tDCS + CIMT: Participants received sham tDCS over the primary motor cortex plus CIMT. The same site and parameters of stimulation were employed, but the stimulator was turned off after 30 seconds of stimulation. This ensured that patients could feel the initial itching sensation at the beginning of tDCS.
Arm/Group | tDCS + CIMT | Sham tDCS + CIMT
Number analyzed (Participants) | 7 | 7
seconds | 68 (34) | 80 (42)

2. Primary Outcome: Cortical Excitability
Description: Motor evoked potential (MEP) Using Transcranial Magnetic Stimulation (TMS), MEP were recorded before and after tDCS (both active and sham).
  The percentage of change in MEP (post versus pre intervention) between the two groups (active and sham) were used for the comparison.
Time Frame: 1 hour
Population: The cortical excitability measurement (MEP) was performed in healthy participants involved in the tDCS+CIMT study (Experiment 2).
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Healthy Participants: Active tDCS + Motor Training | Healthy Participants: Sham tDCS + Motor Training
Number analyzed (Participants) | 20 | 20
percent change | 19.8 (21.4) | 0.8 (8.3)

3. Primary Outcome: Cortical Oscillations - EEG
Description: Recording took place in a dim-lighted room set up with acoustic and electric isolation. EEG was acquired from 64-channels HydroCel Geodesic Sensor Net (Electrical Geodesic Inc., Eugene, OH) and recorded using Net Station running on a MacIntosh G4 computer. Alpha power were used as the main outcome measure. The difference values (e.g., post minus pre tACS) were used for the analysis. The alpha frequency is a brain oscillation that takes place especially when subjects are in a relaxed state, especially eyes closed. In the motor cortex, a decrease in alpha power has been seen during motor performance. Therefore, it could be speculated that a decrease in power in this study would indicate more engagement in motor cortex during the motor performance.
Time Frame: 15 minutes
Population: The brain oscillations measurements were only performed in the tACS study (Experiment 3).
Measure: Mean (Standard Deviation); unit: microVolt^2
Groups:
- Healthy Participants - Active tACS: Subjects will receive 20 min of active tACS
- Healthy Participants - Sham tACS: Subjects will receive 20 min of sham tACS
Arm/Group | Healthy Participants - Active tACS | Healthy Participants - Sham tACS
Number analyzed (Participants) | 7 | 7
microVolt^2 | -0.03 (0.24) | 0.07 (0.16)

ADVERSE EVENTS:
Groups:
- Active tDCS + CIMT - Healthy: subjects will undergo 40 minutes of tDCS at 1mA.
- Sham tDCS + CIMT - Healthy: subjects will undergo 40 minutes of sham tDCS.
- Active tACS - Healthy: Subjects will undergo 20 minutes of active tACS.
- Sham tACS - Healthy: Subjects will undergo 20 minutes of sham tACS.
Arm/Group | tDCS + CIMT - Stroke | Sham tDCS + CIMT - Stroke | Active tDCS + CIMT - Healthy | Sham tDCS + CIMT - Healthy | Active tACS - Healthy | Sham tACS - Healthy
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/10 | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No